CLINICAL TRIAL: NCT05567783
Title: A Double-Blind, Randomized, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy and Safety of VIR-2482 for the Prevention of Illness Due to Influenza A
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of VIR-2482 for the Prevention of Illness Due to Influenza A
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: VIR-2482 1200 mg did not demonstrate efficacy versus placebo in the primary analysis of the primary endpoint
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIR-2482-4002
Record Dates: First submitted 2022-09-24; First posted 2022-10-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Influenza A
Keywords: Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VIR-2482 (Dose 1) (Experimental)
  Interventions: Biological: VIR-2482 (450 mg)
- VIR-2482 (Dose 2) (Experimental)
  Interventions: Biological: VIR-2482 (1200 mg)
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VIR-2482 (450 mg) — VIR-2482 450mg given by intramuscular injection
  Arms: VIR-2482 (Dose 1)
Biological: VIR-2482 (1200 mg) — VIR-2482 1200 mg given by intramuscular injection
  Arms: VIR-2482 (Dose 2)
Biological: Placebo — Sterile 0.9% (w/v) sodium chloride solution given by intramuscular injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of VIR-2482 compared to placebo in preventing influenza A illness in healthy adults 18 to <65 years of age without pre-existing risk factors for serious complications from influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to < 65 years of age, at time of randomization
* Participants must be in good health, determined from medical history and no clinically significant findings from physical examination, 12-lead electrocardiogram (ECG), vital signs, and laboratory values

Exclusion Criteria:

* History or clinical evidence of conditions considered high risk for developing influenza-related complications
* History of confirmed influenza infection within 3 months prior to randomization.
* Febrile illness with or without respiratory symptoms
* History of malignancy within 5 years or participant is under evaluation for malignancy.
* Any condition or receipt of any medication contraindicating IM injection, as judged by the investigator.
* History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis
* Participant has a clinically significant medical condition, physical exam finding, or abnormal laboratory result.
* Prior or planned receipt of any influenza vaccine for the upcoming season.
* Received any investigational agent within 90 days or within 5 half-lives of the investigational agent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2977 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Investigative Site, Anniston, Alabama
  - Investigative Site, Mobile, Alabama
  - Investigative Site, Tempe, Arizona
  - Investigative Site, Long Beach, California
  - Investigative Site, Pomona, California
  - Investigative Site, San Diego, California
  - Investigative Site, Aurora, Colorado
  - Investigative Site, Longmont, Colorado
  - Investigative Site, Fort Myers, Florida
  - Investigative Site, Jupiter, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Pembroke Pines, Florida
  - Investigative Site, Winter Park, Florida
  - Investigative Site, Lilburn, Georgia
  - Investigative Site, Meridian, Idaho
  - Investigative Site, Chicago, Illinois
  - Investigative Site, South Bend, Indiana
  - Investigative Site, El Dorado, Kansas
  - Investigative Site, Lenexa, Kansas
  - Investigative Site, Wichita, Kansas
  - Investigative Site, Lexington, Kentucky
  - Investigative Site, Versailles, Kentucky
  - Investigative Site, Metairie, Louisiana
  - Investigative Site, New Orleans, Louisiana
  - Investigative Site, Methuen, Massachusetts
  - Investigative Site, Kansas City, Missouri
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, Rochester, New York
  - Investigative Site, Monroe, North Carolina
  - Investigative Site, Raleigh, North Carolina
  - Investigative Site, Cincinnati, Ohio
  - Investigative Site, Edmond, Oklahoma
  - Investigative Site, Yukon, Oklahoma
  - Investigative Site, Anderson, South Carolina
  - Investigative Site, North Charleston, South Carolina
  - Investigative Site, Spartanburg, South Carolina
  - Investigative Site, Rapid City, South Dakota
  - Investigative Site, Elizabethton, Tennessee
  - Investigative Site, Knoxville, Tennessee
  - Investigative Site, Austin, Texas
  - Investigative Site, Cedar Park, Texas
  - Investigative Site, Dallas, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, San Angelo, Texas
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Tomball, Texas
  - Investigative Site, Layton, Utah
  - Investigative Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tan SK, Cebrik D, Plotnik D, Agostini ML, Boundy K, Hebner CM, Yeh WW, Pang PS, Moya J, Fogarty C, Darani M, Hayden FG. A Randomized, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of VIR-2482 in Healthy Adults for Prevention of Influenza A Illness (PENINSULA). Clin Infect Dis. 2024 Oct 15;79(4):1054-1061. doi: 10.1093/cid/ciae368. PMID 39036981

RESULTS

PARTICIPANT FLOW:
Groups:
- VIR-2482 (450 mg): VIR-2482 (450 mg): VIR-2482 450 mg given by intramuscular injection
Period: Overall Study
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Started | 989 | 995 | 993
Received Study Intervention | 981 | 992 | 983
Completed | 0 | 0 | 0
Not Completed | 989 | 995 | 993
Not completed — Death | 2 | 3 | 0
Not completed — Lost to Follow-up | 25 | 19 | 17
Not completed — Physician Decision | 10 | 7 | 9
Not completed — Study Terminated by Sponsor | 924 | 937 | 941
Not completed — Withdrawal by Subject | 23 | 27 | 24
Not completed — Incarcerated | 1 | 0 | 0
Not completed — Participant randomized in error | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received any amount of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo | Total
Number analyzed (Participants) | 981 | 992 | 983 | 2956
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (12.52) | 39.6 (11.73) | 39.7 (12.29) | 39.5 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 545 | 523 | 530 | 1598
  Male | 436 | 469 | 453 | 1358
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 371 | 369 | 357 | 1097
  Not Hispanic or Latino | 606 | 622 | 620 | 1848
  Unknown or Not Reported | 4 | 1 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 7 | 7 | 21
  Asian | 26 | 29 | 26 | 81
  Native Hawaiian or Other Pacific Islander | 5 | 4 | 4 | 13
  Black or African American | 154 | 176 | 166 | 496
  White | 752 | 747 | 758 | 2257
  More than one race | 17 | 11 | 6 | 34
  Unknown or Not Reported | 20 | 18 | 16 | 54
Region of Enrollment [Number; unit: participants]
  United States | 981 | 992 | 983 | 2956
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index at Screening
  kg/m^2 | 27.34 (4.085) | 27.44 (4.167) | 27.4 (4.071) | 27.34 (4.107)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Protocol-defined Influenza-like Illness (ILI) With Confirmed Influenza A (by Reverse Transcription Polymerase Chain Reaction [RT-PCR])
Description: Protocol-defined ILI with confirmed influenza A defined as RT-PCR confirmed influenza A with at least one respiratory symptom and at least one systemic symptom
Time Frame: Up to 24 Weeks
Population: Full Analysis Set (all randomized who did not have confirmed influenza infection within 3 months prior to randomization, did not receive an influenza vaccination for the upcoming influenza season, and received any amount of study intervention). Participants were analyzed according to the randomized study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
percentage of participants | 2.45 | 2.12 | 2.54
Statistical Analysis 1: Comparison: VIR-2482 (1200 mg) vs Placebo; Test type: Superiority; p = 0.5552, Poisson regression — two-sided, alpha=0.05; Estimated using Poisson regression of multiple imputed data with treatment group the only factor in the model; Relative risk reduction (RRR, %) = 15.85, 95% CI 2-sided [-49.27 to 52.56] — RRR and 95% CI estimated using Poisson regression of multiple imputed data with treatment group was the only factor in the model
Statistical Analysis 2: Comparison: VIR-2482 (450 mg) vs Placebo; Test type: Superiority; Relative risk reduction (RRR, %) = 3.78, 95% CI 2-sided [-67.23 to 44.63] — RRR and 95% CI estimated using Poisson regression of multiple imputed data with treatment group the only factor in the model; 95% CI are nominal and not adjusted for multiple comparisons

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Up to 26 Weeks
Population: Participants who received any amount of study intervention. Participants were analyzed according to study intervention received.
Measure: Count of Participants; unit: Participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
Participants | 636 | 613 | 639

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Time Frame: Up to 26 Weeks
Population: Participants who received any amount of study intervention. Participants were analyzed according to the study intervention received.
Measure: Count of Participants; unit: Participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
Participants | 10 | 13 | 9

4. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: AESI is anaphylaxis per MedDRA anaphylaxis algorithmic SMQ
Time Frame: Up to 26 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Defined as a graded abnormality in systolic blood pressure, diastolic blood pressure, pulse, respiratory rate, or oral temperature as per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials at any time on/after receipt of study intervention.
Time Frame: Up to 26 Weeks
Population: Participants who received any amount of study intervention and had a post-baseline vital sign measurement. Participants were analyzed according to the study intervention received.
Measure: Count of Participants; unit: Participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 981
Participants | 678 | 662 | 648

6. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Defined as graded abnormality in chemistry, hematology, liver function, or urinalysis clinical laboratory values as per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Trials at any time on/after receipt of study intervention.
Time Frame: Up to 26 Weeks
Population: Participants who received any amount of study intervention and had a post-baseline clinical laboratory assessment. Participants were analyzed according to the study intervention received.
Measure: Count of Participants; unit: Participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 978 | 988 | 976
Participants | 961 | 971 | 961

7. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: Injection site reactions from the study intervention diary card
Time Frame: Up to Day 7 following study intervention administration
Population: Participants who received any amount of study intervention . Participants were analyzed according to the study intervention received.
Measure: Count of Participants; unit: Participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
Participants
  Any injection site reaction | 292 | 293 | 272
  Pain | 279 | 277 | 260
  Erythema | 7 | 10 | 5
  Induration | 8 | 12 | 3
  Swelling | 10 | 13 | 2
  Bruising | 17 | 20 | 21

8. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: Systemic reactions from the study intervention diary card
Time Frame: Up to Day 7 following study intervention administration
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
Participants
  Any systemic reaction | 265 | 283 | 268
  Headache | 160 | 168 | 175
  Myalgia | 135 | 169 | 149
  Malaise | 117 | 130 | 123
  Shivering | 44 | 60 | 43
  Fever | 11 | 11 | 13

9. Secondary Outcome: Percentage of Participants With CDC-defined Influenza-like Illness (ILI) With Confirmed Influenza A (by Reverse Transcription Polymerase Chain Reaction [RT-PCR])
Description: CDC-defined ILI with RT-PCR confirmed influenza A
Time Frame: Up to 24 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
percentage of participants | 1.53 | 0.71 | 1.73
Statistical Analysis 1: Comparison: VIR-2482 (1200 mg); Test type: Superiority; Relative risk reduction (RRR, %) = 57.23, 95% CI 2-sided [-2.51 to 82.15] — RRR and 95% CI estimated using Poisson regression of multiple imputed data with treatment group the only factor in the model; 95%CI are nominal and not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: VIR-2482 (450 mg) vs Placebo; Test type: Superiority; Relative risk reduction (RRR, %) = 11.45, 95% CI 2-sided [-76.25 to 55.51] — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Percentage of Participants With WHO-defined Influenza-like Illness (ILI) With Confirmed Influenza A (by Reverse Transcription Polymerase Chain Reaction [RT-PCR])
Description: WHO-defined ILI with RT-PCR confirmed influenza A
Time Frame: Up to 24 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
Number analyzed (Participants) | 981 | 992 | 983
percentage of participants | 1.22 | 0.6 | 1.12
Statistical Analysis 1: Comparison: VIR-2482 (1200 mg) vs Placebo; Test type: Superiority; Relative risk reduction (RRR, %) = 44.13, 95% CI 2-sided [-50.49 to 79.26] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: VIR-2482 (450 mg) vs Placebo; Test type: Superiority; Relative risk reduction (RRR, %) = -9.80, 95% CI 2-sided [-147.41 to 51.27] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: through study completion for each participant, up to approximately 43 weeks
Arm/Group | VIR-2482 (450 mg) | VIR-2482 (1200 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/981 | 3/992 | 0/983
Serious Adverse Events (participants affected / at risk) | 10/981 | 13/992 | 9/983
Other Adverse Events (participants affected / at risk) | 454/981 | 450/992 | 460/983
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIR-2482 (450 mg) (N=981) | VIR-2482 (1200 mg) (N=992) | Placebo (N=983)
Appendicitis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Schizoaffective disorder bipolar type (Psychiatric disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Uterine malposition (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic organ prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 — General disorders and administration site conditions
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIR-2482 (450 mg) (N=981) | VIR-2482 (1200 mg) (N=992) | Placebo (N=983)
Upper respiratory tract infection (Infections and infestations) | 243 | 245 | 248
COVID-19 (Infections and infestations) | 93 | 91 | 106
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 95 | 87 | 75
Cough (Respiratory, thoracic and mediastinal disorders) | 88 | 84 | 72
Viral infection (Infections and infestations) | 56 | 48 | 70
Myalgia (Musculoskeletal and connective tissue disorders) | 51 | 36 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT05567783/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT05567783/SAP_001.pdf